CLINICAL TRIAL: NCT05256511
Title: Incidence of Ventilator-associated Lower Respiratory Tract Infections Among Patients With SARS-CoV-2 Infection Throughout the First and the Second Wave of the Pandemic: a European Comparative Cohort Study
Brief Title: COVID-19 and VA-LRTI: Second Versus First Wave of the Pandemic
Acronym: CoVAPid2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: HLJ_2022_01
Record Dates: First submitted 2022-02-24; First posted 2022-02-25 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-02

CONDITIONS: Severe COVID-19
Keywords: SARS-CoV-2; ventilator-associated tracheobronchitis; ventilator-associated pneumonia; bacterial co-infection; COVID-associated pulmonary aspergillosis
MeSH Terms: conditions — COVID-19; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 first wave: Patients with confirmed SARS-CoV-2 infection and receiving invasive mechanical ventilation for more than 48h, in the first wave of the pandemic, starting on 01-01-2020
- SARS-CoV-2 second wave: Patients with confirmed SARS-CoV-2 infection and receiving invasive mechanical ventilation for more than 48h, in the second wave of the pandemic, starting on 10-01-2020

SUMMARY:
Multicenter observational retrospective cohort study aiming at comparing the incidence of ventilator-associated lower respiratory tract infections between COVID-19 patients from the first and the second wave of the pandemic.

DETAILED DESCRIPTION:
CoVAPid2 is a multicenter retrospective observational cohort study aiming at comparing the incidence of ventilator-associated lower respiratory tract infections between COVID-19 patients from the first and the second wave of the pandemic. Patients with confirmed SARS-CoV-2 community-acquired pneumonia and receiving invasive mechanical ventilation for more than 48h in the participating ICUs from the start of COVID pandemic are eligible for this study. Consecutive patients will be included from the beginning of the first wave (starting on 01-01-2020, data already collected in the CoVAPid1 study) and the second wave (starting on 10-01-2020). 10-20 patients per wave will be included in each center. VAT and VAP are defined using clinical, radiological and quantitative microbiological criteria.

ELIGIBILITY:
Inclusion Criteria:

* Major (18 years and older)
* Admitted to the ICU
* Intubated and mechanically ventilated for more than 48 hours
* With a confirmed community-acquired SARS-CoV2 pneumonia

Exclusion Criteria:

* Refusal to participate
* Lack of social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed SARS-CoV-2 community-acquired pneumonia and receiving invasive mechanical ventilation for more than 48h in the participating ICUs from the start of COVID pandemic are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 1136 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of ventilator-associated lower respiratory tract infection (ventilator-associated pneumonia and ventilator associated tracheobronchitis) | from day 3 of mechanical ventilation to extubation or day 28 post-intubation

SECONDARY OUTCOMES:
Cumulative incidence of ventilator-associated tracheobronchitis | from day 3 of mechanical ventilation to extubation or day 28 post-intubation
Cumulative incidence of ventilator-associated pneumonia | from day 3 of mechanical ventilation to extubation or day 28 post-intubation
Prevalence of early bacterial coinfection | from day 0 to day 2 of mechanical ventilation
Cumulative incidence of COVID-associated pulmonary aspergillosis | from day 3 of mechanical ventilation to extubation or day 28 post-intubation
ICU mortality | at day 28
Mortality | at day 28
Duration of mechanical ventilation (number of days under mechanical ventilation) | from the start of mechanical ventilation to extubation or day 28 after intubation
Duration of ICU stay (number of days in the ICU) | from the ICU admission to discharge or day 28 after admission

CONTACTS AND LOCATIONS:
Overall Officials: Saad NSEIR, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Salengro - Hopital B Chr Lille, Lille, France